CLINICAL TRIAL: NCT04778696
Title: PASO - Automated Template Matching for PVC Ablation: A Randomised Clinical Trial
Brief Title: PASO Automated Template Matching for PVC Ablation
Acronym: PAsT-PVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKK-PASTPVC-2018
Record Dates: First submitted 2018-02-16; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: PVC - Premature Ventricular Complex; Cardiomyopathies; Heart Failure; Ventricular Tachycardia
MeSH Terms: conditions — Ventricular Premature Complexes; Cardiomyopathies; Heart Failure; Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: 1:1 simple randomisation
Who Masked: Participant, Investigator
Masking Description: Patients will be masked to treatment arm. Investigator performing statistical analysis and adjudicating outcomes will be masked to treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional pace mapping (Active Comparator): Conventional PVC pace mapping without visual guidance of PASO
  Interventions: Procedure: Conventional Pacemapping
- PASO pace mapping (Experimental): PASO pace mapping with visualisation in CARTO3
  Interventions: Procedure: PASO Pacemapping

INTERVENTIONS:
Procedure: PASO Pacemapping — Using the PASO pacemapping visualisation module of CARTO3
  Arms: PASO pace mapping
Procedure: Conventional Pacemapping — without visualisation in 3D mapping
  Arms: conventional pace mapping

SUMMARY:
Pacemapping is an essential tool during ablation of idiopathic PVC and VT. Automated template matching has been shown to have a significant influence on PVC ablation procedures, but the PASO module of CARTO3 has not been studied in a randomized trial. The Aim of this study is to evaluate the additional benefit of PASO template matching on PVC ablation procedure with regard to procedural parameters and outcome when compared with conventional pace mapping. A total of 144 pts will be randomised in a 1:1 fashion to PVC ablation guided by conventional pacemapping vs PVC ablation guided by PASO pacemapping. Patients will be follow up with Holter-ECG and TTE after 3 and 12 months.

DETAILED DESCRIPTION:
Introduction / Rationale Premature ventricular contractions (PVC) in the otherwise healthy heart are not associated with increased mortality in the absence of a short coupling interval or a compromised left ventricular function and do not require treatment if asymptomatic . Symptomatic idiopathic PVC or VT on the other hand can burden patients with recurring palpitations, dizziness, dyspnea and possibly syncope in cases of fast VT. A reversible decrease in left ventricular function as a result of a high PVC burden has been reported even in patients with no underlying cardiomyopathy . Radiofrequency Ablation (RFA) is a well-established method to treat idiopathic PVC and VT, and is associated with satisfying long-term results. Pacemapping is an essential tool during ablation of idiopathic PVC and VT. Automated template matching has been shown to have a significant influence on PVC ablation procedures, but the PASO module of CARTO3 has not been studied in a randomized trial.

Aim of the study To evaluate the additional benefit of PASO template matching on PVC ablation procedure with regard to procedural parameters and outcome when compared with conventional pace mapping.

Hypothesis PASO guidance during PVC / VT ablation has a significant impact on outcome after catheter ablation of idiopathic PVC / VT.

Study design This study is planned as a two-center trial. All patients presenting for de novo ablation of idiopathic ventricular arrhythmia will be included and randomized in a 1:1 fashion in this open-label, two-center, randomized controlled trial.

In patients randomized to the PASO / intervention group pacemapping will be guided by automated template matching of the PASO module of CARTO3.

In patients randomized to the conventional / control group conventional pacemapping will be employed.

A 3D electroanatomic geometry including activation mapping will be acquired in all patients using CARTO3. Sedation, catheters and monitoring during and after CA, will not differ from standard clinical practice and will be the same for both groups.

Follow-up after 3 and 12 months will assess PVC burden by Holter ECG, symptoms through a standardized questionnaire and LV function by TTE

Duration and study size Based on prior findings ("Impact of Automated Template Matching during PVC Ablation: Results from a Randomized Controlled Trial" Lüker et al. ESC 2014 poster presentation) 144 pts have to be randomized to detect a significant difference with respect to ablation success at follow-up (alpha 0.05, power 80%).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed, written consent
* ventricular arrhythmia (PVC or VT) with indication for CA

Exclusion Criteria:

* Patients under guardianship or with mental disorders / disabilities
* Polymorphic PVC / VT
* ongoing myocardial ischaemia
* pregnancy
* valve replacement that prevents access to the suspected site of PVC origin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
PVC recurrence in Holter ECG | 12 weeks after ablation procedure
  Assessment of PVC as % of total number heart beats in a 24 hours Holter ECG

SECONDARY OUTCOMES:
Symptomatic recurrence | between 3 and 12 months after ablation
  recurrence of PVC according to the patients symptoms
LV ejection fraction assessment (%) | between 3 months and 12 months after ablation
  Change in LV ejection fraction after ablation (%)
Procedure duration | From groin puncture to sheath removal
  Procedure duration (min)
Prcedural fluoroscopy parameters | From groin puncture to sheath removal
  Fluoroscopy dose (Gy x cm2) and time (min)
Procedural ablation parameters | From groin puncture to sheath removal
  Number of RF lesions (n) and acute ablation success (cessation of PVC)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No